CLINICAL TRIAL: NCT02303197
Title: A Randomized,Controlled Clinical Trial on the Efficacy and Safety of Chining Decoction in the Treatment of Radiation Stomatitis.
Brief Title: Clinical Trial on the Efficacy and Safety of Chining Decoction in the Treatment of Radiation Stomatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TianjinCIH
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2014-10

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; chemoradiotherapy; radioactive stomatitis
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ChiNing decoction (Experimental): 60ml ChiNing decoction by mouth，three times a day for 46 days.
  Interventions: Drug: ChiNing decoction
- rhEGF spray (No Intervention): The rhEGF spray spray on the oral mucosal surface irradiated area, 3 times a day for 46 days.

INTERVENTIONS:
Drug: ChiNing decoction — ChiNing decotion was reformed by Liangge San that was stemed from Prescriptions of the Bureau of Taiping People.
  Other Names: Addition and subtraction of Liangge San
  Arms: ChiNing decoction

SUMMARY:
This study evaluates the efficiency and safety of ChiNing decoction to head and neck cancer patients with radioactive stomatitis. Half of participants will receive ChiNing decoction, while others will receive recombinant human epidermal growth factor (rhEGF) spray.

DETAILED DESCRIPTION:
This study uses randomized, controlled clinical research methods, through the observation of the treatment group (ChiNing decoction orally) and control group (recombinant human epidermal growth factor rhEGF spray on oral mucosal surface ) at different time points before and after radiotherapy, to evaluate the radiotherapy of acute radiation oral mucosa reaction (RTOG grade), quality of life score (EORTCQLQ-H&N35 scale), oral pain (VAS score) and patient body weight changes of the two groups. At the same time，this study takes cast-off cells of oral mucosal to observe the microscopic characteristics of oral mucosa, and uses the ELISA method to detect IL-6 and TNF- alpha content in the saliva before and after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients with pathology and / or cytologic diagnosis;
* Age 18~75 years old;
* The expected life is more than 3 months;
* The Karnofsky score (Karnofsky) ≥70 points;
* The first course of radiotherapy in patients;
* Patients had not received any anti tumour therapies for example of operation, radiotherapy,chemotherapy, biological treatment or isotope therapy system;
* Patients volunteered to participate in this test and signed the informed consent, understand the purpose and test steps of the test, good compliance, comply with the relevant requirements of this test scheme;
* No history of oral ulcer and salivary gland diseases

Exclusion Criteria:

* That do not meet the above the inclusion criteria;
* Advanced critical cases, the expected survival is less than 3 months;
* The patients had serious complications, such as cachexia, hepatic encephalopathy, gastrointestinal bleeding and coagulation functionobstruction, su ch as abnormal;
* The submandibular gland pathological changes;
* During radiotherapy taking other drugs in patients with treatment of stomatitis;
* The patients with serious heart, brain, liver, kidney function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Grading standard of RTOG in acute radiation injury of oral mucosal | 8 days
  Score before the radiotherapy and every 1 week after the begining of the radiotherapy and after the end of radiotherapy

SECONDARY OUTCOMES:
The visual analogue scale of oral pain | 8 days
  Score before the radiotherapy and every 1 week after the begining of the radiotherapy and after the end of radiotherapy
EORTCQLQ-H&N35 | 8 days
  Score before the radiotherapy and every 1 week after the begining of the radiotherapy and after the end of radiotherapy
patient body weight changes | 8 days
  Score before the radiotherapy and every 1 week after the begining of the radiotherapy and after the end of radiotherapy
Safety index | 2 days
  Chech the blood routine, urine routine, liver and kidney function, electrocardiogram before and after the radiotherapy

OTHER OUTCOMES:
IL-6 and TNF- alpha content | 2 days
  With distilled water repeatedly rinse of 1 min, 10 min after discarding the first mouthful of saliva, sit down, spit saliva to the sterile tube in 4 Centigrade， before and after the radiotherapy
takes cast-off cells of oral mucosal | 2 days
  rinse the mouth with the physiological salt water , scrap sides of buccal oral mucosa 2 times appropriate efforts with appropriate effort, painted on a slide，before and after the radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Cong Wang, Master, Principal Investigator — National Clinical Research Center for Cancer of China
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Ryu SH, Kang KM, Moon SY, Chai GY, Hong JP, Cho KO, Kang MI, Choi EK, Lee SW. Therapeutic effects of recombinant human epidermal growth factor (rhEGF) in a murine model of concurrent chemo- and radiotherapy-induced oral mucositis. J Radiat Res. 2010;51(5):595-601. doi: 10.1269/jrr.10069. PMID 20921827
- [Background] Spielberger R. Current management of oral mucositis. Clin Adv Hematol Oncol. 2005 Oct;3(10):769-71. No abstract available. PMID 16258486
- [Background] Wang B, Cao SH, Wang YQ. [Effects of modified liangge powder contained serum on LPS stimulated TLR4 expression and release of cytokines in mouse platelets]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 2012 May;32(5):681-4. Chinese. PMID 22679734
- [Background] Yu LZ, Jiang AD, Cheng YY, Lin H, Qin QH, Ma XD. [Liangge san effects the expression of CD14 and scaverger receptor in the Kupffer cells of liver of endotoxemia mice]. Zhongguo Zhong Yao Za Zhi. 2006 Feb;31(3):220-3. Chinese. PMID 16573003
- [Background] Jiang AD, Yu LZ, Gong XW, Deng P, Ma XD. [Effect of Liangge San on lipopolysaccharide-induced nuclear factor kappa B activation in cultured mouse macrophages]. Di Yi Jun Yi Da Xue Xue Bao. 2005 Jun;25(6):619-22. Chinese. PMID 15958292